CLINICAL TRIAL: NCT03459872
Title: Acupuncture Outcomes Based Rehabilitation Through Measurement of Fine Motor Control
Brief Title: Acupuncture Outcomes Based Rehabilitation
Status: Completed | Type: Observational
Sponsor: Community Medical Foundation for Patient Safety (Other)
Collaborators: Red Oak Instruments, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: RU-Fit Acu 1
Record Dates: First submitted 2018-02-26; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Pain
Keywords: acupuncture; quantitative data; outcomes based rehabilitation; fine motor control
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Acupuncture Intervention group: RU-Fit gathers measurements of fine motor control were gathered from this group before and after acupuncture treatments.
  Interventions: Procedure: Acupuncture; Device: RU-Fit
- Control/ Non-Intervention: This group received no intervention but still had measurements of fine motor control gathered from RU-Fit medical device.
  Interventions: Device: RU-Fit

INTERVENTIONS:
Procedure: Acupuncture — Alternative medicine therapeutic intervention
  Groups: Acupuncture Intervention group
Device: RU-Fit — FDA approved medical device for the measurement of fine motor control

SUMMARY:
Can acupuncture be quantified. This study sets out to observe if there are measurable effects of fine motor control that are attributable to acupuncture. The study utilizes an FDA approved medical device for measurements of fine motor control called the RU-Fit.

DETAILED DESCRIPTION:
Context: Currently there is a high demand for evidence-based research in the field of Acupuncture. The medical practice of acupuncture has existed for thousands of years and purportedly has been successful at managing a wide array of health conditions. Producing objective/quantitative data that rule out any possibility of placebo effect has proved burdensome.

Objectives: This exploratory study seeks to determine if physiological measurements of fine motor control can be changed after receiving an acupuncture treatment. Can this change demonstrate the effectiveness of the treatment? Design, Setting, Participants, Interventions: This study looked at acupuncture patients undergoing treatments for pain relief, and general minor injury to determine whether or not observable changes could be detected in the fine motor control of the hands after acupuncture treatments.

Two groups of 50 subjects were used in the study. The test group was given a fine motor control test prior to and after their acupuncture therapy to determine if any changes could be measured.

The control group was given two fine motor control tests without acupuncture treatment with a 40 minute delay between the tests to replicate the test group timing. This study was conducted at a non-profit community clinic between the dates of 9/28/16 & 2/19/17.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 13 years old or older
* Study participants were selected from the acupuncture patient population freely visiting the clinic. Patients were asked if they would be interested in a research study. They were informed about the objectives of the study, what their role would be and that this was a free non-invasive test that they would undergo before and after their regular acupuncture treatment. Before inclusion into the program, patients are provided with informed consent forms and after agreeing and signing the form, individuals then become participants.

Exclusion Criteria:

* Younger than 13 years old

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants were selected from the acupuncture patient population freely visiting the clinic. Patients were asked if they would be interested in a research study. They were informed about the objectives of the study, what their role would be and that this was a free non-invasive test that they would undergo before and after their regular acupuncture treatment. Before inclusion into the program, patients are provided with informed consent forms and after agreeing and signing the form, individuals then become participants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2017-01-21 (Actual); Study Completion 2017-02-19 (Actual)

PRIMARY OUTCOMES:
Assessing Changes in Fine Motor Control from Acupuncture | Before and after acupuncture treatment or space of 40 minutes for control group between testing
  Fine Motor Control measurements (probability percentage of normal capability) from RU-Fit, FDA approved medical device

IPD SHARING:
Plan to Share IPD: No
Information will be shared regarding measurements that were obtained from medical device testing such as fine motor control